CLINICAL TRIAL: NCT05398094
Title: Phase II Clinical Trial of AMG510 (Sotorasib) in Stage III Unresectable NSCLC KRAS p.G12C Patients and Medically Ineligible for Concurrent Chemo-radiotherapy
Brief Title: Clinical Trial of AMG510 in Stage III Unresectable NSCLC KRAS p.G12C Patients and Ineligible for Chemo-radiotherapy
Acronym: MERIT-lung
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 20/10_MERIT-lung; 2021-004576-34 (EudraCT Number)
Record Dates: First submitted 2022-05-13; First posted 2022-05-31 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer Stage III; KRAS P.G12C
Keywords: Sotorasib; Unresectable; Chemo-radiotherapy; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Induction treatment + Post-Induction Phase (Experimental): Patients enrolled in the study will receive AMG510 (Sotorasib) 960mg once daily for 2 cycles (Q4W) in the induction phase and AMG510 (Sotorasib) 960 mg once daily (Q4W) in the treatment postinduction phase.
  Treatment post-induction phase only for patients with SD, PR or CR after induction treatment. This treatment will be administered until progression disease (PD), unacceptable toxicity, patient or physician's decision to discontinue or death.
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — AMG510 (Sotorasib) is small molecule that specifically and irreversibly inhibits the KRAS-G12C mutant protein. AMG510 (Sotorasib) finished product is presented as tablets containing 120mg and will be packaged in bottles of 120 tablets.
  Other Names: AMG510

SUMMARY:
Open-label, non-randomised, exploratory, phase II, multi-centre clinical trial. 43 unresectable stage III (IIIA-N2, IIIB, IIIC) KRAS p.G12C non-small cell lung cancer patients will be enrolled in this trial to evaluate the efficacy of induction treatment of AMG510 (Sotorasib) plus AMG510 (Sotorasib) treatment post-induction as measured by Progression Free Survival at 12 months.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, exploratory, phase II multi-centre clinical trial.The total sample size is 43 patients. The population to be included are unresectable stage III (IIIA-N2, IIIB, IIIC) KRAS p.G12C non-small cell lung cancer patients.

Patients randomised will receive AMG510 (Sotorasib) 960mg once daily for 2 cycles (Q4W) in the induction phase and AMG510 (Sotorasib) 960 mg once daily (Q4W) in the treatment post-induction phase. Treatment post-induction phase only for patients with SD, PR or CR after induction treatment. This treatment will be administered until progression disease (PD), unacceptable toxicity, patient or physician's decision to discontinue or death.

The primary objective is to assess the efficacy of induction treatment of AMG510 (Sotorasib) plus AMG510 (Sotorasib) treatment post-induction as measured by Progression Free Survival at 12 (PFS12) months according to Response Evaluation Criteria in Solid Tumors (RECIST) version PFS are defined as the time from inclusion until objective tumor progression or death.

Patient accrual is expected to be completed within 5 years and a half, treatment is planned to extend for 1.5 years and the patients will be followed up for 2 years. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, aged ≤ 80 years old
* 2. ECOG performance status of 0-1
* 3. Histologically or cytologically confirmed, unresectable Stage III (IIIA-N2, IIIB and IIIC) NSCLC according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology.
* 4. Patients who have documentation of KRAS p.G12C prior to enrollment. This determination can be done either by solid or liquid biopsy.
* 5. No prior treatment for unresectable Stage III (IIIA-N2, IIIB and IIIC) NSCLC.
* 6. Having a life expectancy ≥ 12 weeks
* 7. Patients must be ineligible for concurrent chemo-radiotherapy because of:

  1. Tumor size ≥ 5 cm and lymph node N2 involvement
  2. The target lesion has to be bulky disease and/or more than 35% of the total volume of the two lungs should receive more than 20 Gy (V20) or inadequate pulmonary function
  3. Interstitial Lung diseases
  4. Prior treatment with thoracic radiotherapy for any reason
  5. Or under decision of a tumor committee as inappropriate due to local characteristics to perform treatment upfront
* 8. PET-CT at baseline is mandatory to confirm the absence of distant disease and to confirm unresectable disease
* 9. PET-CT positive mediastinic adenopathies must be histologically confirmed. Mediastinic involvement could be considered without histological test when no margin can be distinguished in the lymph node mass.
* 10. Brain CT or MRI is mandatory
* 11. Patients with at least 1 measurable lesion, as defined by RECIST v1.1.
* 12. Adequate hematologic and organ function.
* 13. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention.
* 14. Willingness and ability to comply with scheduled visits and study procedures
* 15. For female patients of childbearing potential, a negative pregnancy test must have been documented prior to enrollment (within 14 days prior to enrollment).
* 16. For female patients of childbearing potential, agreement (by patient and/or partner) to usea highly effective form(s) of contraception that results in a low failure rate (< 1% per year)when used consistently and correctly, and to continue its use for 7 days after the last dose of AMG510 (Sotorasib). No hormonal methods and preferably barrier method always containing a spermicide, intrauterine device (IUD): intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
* 17. For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate [< 1% per year] when used consistently and correctly, and to continue its use for 7 days after the last dose of AMG510 (Sotorasib).
* 18. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to enrollment.
* 19. QTc interval must be ≤ 470 msec in females and ≤ 450 msec in males, based on the average obtained from three ECG.

Exclusion Criteria:

* 1. Patients with a known sensitizing mutation in the epidermal growth factor receptor (EGFR) gene, ALK translocations or ROS1 mutations
* 2. Weight loss >10% within the previous 3 months
* 3. Patients with uncontrolled neuropathy (sensory) grade 2 or greater regardless of cause according to CTCAE v5.0
* 4. Major surgery within 28 days of study day 1
* 5. Significant gastrointestinal disorder that results in significant malabsorption, requirement for intravenous alimentation, or inability to take oral medication
* 6. Significant cardiovascular disease, such as New York Heart Association cardiac disease (ClassII or greater), myocardial infarction within 6 months prior to study day 1, unstable arrhythmias or unstable angina
* 7. Ongoing cardiac dysrhythmias of CTCAE grade ≥2, uncontrolled atrial fibrillation of any grade or QTcF interval > 470ms
* 8. Severe infections within 4 weeks prior to randomization including, but not limited to hospitalization for complications of infection, bacteremia or severe pneumonia
* 9. Therapeutic oral or intravenous antibiotics within 2 weeks prior to randomization
* 10. Patients with any concomitant and uncontrolled medical disorder
* 11. Patients with vena cava syndrome
* 12. Malignant pleural or pericardial effusion: both will be considered as suggestive of metastaticdisease. Also, are excluded those with negative cytology but being exudates. Patients with non-visible by thoracic X-ray pleural effusion or too small to be safely punctured could be included.
* 13. Prior treatment with anti-neoplasic drugs
* 14. Malignancies other than NSCLC within 3 years prior to enrollment
* 15. Women who are pregnant, lactating, or intending to become pregnant during the study.
* 16. Positive test for HIV. All patients will be tested for HIV prior to inclusion into the study; patients who test positive for HIV will be excluded from the clinical study.
* 17. Patients with active hepatitis B or hepatitis C.
* 18. Active tuberculosis.
* 19. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.
* 20. Patients with illnesses or conditions that interfere with their capacity to understand follow and/or comply with study procedures.
* 21. Known or suspected hypersensitivity to drugs with similar chemical structures to the study drug
* 22. Evidence of any other disorder or significant laboratory finding that makes the patient undesirable to participate in the study
* 23. Use of strong inducers of CYP3A4 within 14 days of half-lives (whichever is longer) prior to study day 1
* 24. Use of proton pump inhibitors within 14 days to study day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the treatment in terms of the Progression Free Survival (PFS) | From the date of first dose of induction treatment until 6 months
  PFS defined as the length of time from the date of end of post-induction treatment to the date of the first documented progression of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Overall response rate (ORR) of AMG510 (Sotorasib) | From the date of the end of treatment until 12 months and 24 months
  Overall response will be assessed per RECIST v1.1 criterion. ORR is defined as the proportion of patients who have a partial or complete response to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity.
Overall Survival (OS) rate of treatment with AMG510 (Sotorasib) | From the date of the start of treatment until 12 and 24 months
  OS defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
Detect and collect the sites of first failure | From the date of the start of treatment until the date of last follow up, assessed up to 24 months
  Sites of the first failure defined as the first site of the body of documented relapse or progression of the lung cancer disease after a period of improvement.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the subject written informed consent signature to 30 days from last dose of treatment.
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — Fundación GECP President
Locations (20):
- Spain (20):
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital de Son Espases, Palma de Mallorca, Mallorca
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Parc Taulí, Barcelona
  - Hospital De Basurto, Bilbao
  - ICO Girona, Hospital Josep Trueta, Girona
  - Hospital Clínico San Cecilio De Granada, Granada
  - Complejo Hospitalario De Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitari Son Llatzer, Palma de Mallorca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital General Universitario De Valencia, Valencia
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org